CLINICAL TRIAL: NCT01658748
Title: A Pilot Study to Examine Deep Brain Stimulation (DBS) in the Basolateral Nucleus (BLn) of the Amygdala for the Management of Symptoms in Veterans With Chronic and Treatment-Refractory Combat-related Post-Traumatic Stress Disorder (PTSD)
Brief Title: A Pilot Study of Deep Brain Stimulation of the Amygdala for Treatment-Refractory Combat Post-Traumatic Stress Disorder
Acronym: ADIP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not finalized
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N1112-I; 1/01RX001112-01 (Other Grant/Funding Number: Department of Veterans Affairs); PCC-2012 (Other: VA Greater Los Angeles Healthcare System)
Record Dates: First submitted 2012-07-28; First posted 2012-08-07 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Pilot Study; Longitudinal Study; Amygdaloid Body; Insula of Reil; Cortex, prefrontal; Stimulation, Deep Brain; Chronic Post Traumatic Stress Disorder; Combat Stress Disorder; Social Adjustments; Positron-Emission Tomography, Computed Tomography
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders; Social Adjustment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Week 0 Medtronic 3387 electrodes/Activa PC amygdala DBS (Active Comparator): Patients randomized to this arm will have stimulators turned on approximately 1 week after the 3-4 week post-surgery EEG telemetry session that determines safety parameters for stimulator settings. Subjects will be followed weekly for the next 12 weeks, with adjustments in stimulator settings according to prescribed protocol based on changes in rating scale scores (CAPS, CGI-I, ADIPS, LFIPS, HAMA, MADRS, YMRS).
  Interventions: Device: Week 0 Medtronic 3387 electrodes/Activa PC amygdala DBS; Device: Week 12 Medtronic 3387 electrodes/Activa PC amygdala DBS
- Week 12 Medtronic 3387 electrodes/Activa PC amygdala DBS (Sham Comparator): Patients randomized to this arm will undergo the same procedures and same visit frequency as those in the week 0 stimulation arm, except that the actual stimulation settings will be kept at 0 V, 0 Hz, and the patient, study psychiatrist who does the ratings, and study neurosurgeon who does neurological clinical assessments will be blind to whether the subject is receiving actual or sham stimulation. Only the study neurophysiologist will know whether the patient is in the active or sham stimulation arm during these 12 weeks. After week 12, subjects in this week will begin to receive active stimulation according to pre-specified protocol.
  Interventions: Device: Week 12 Medtronic 3387 electrodes/Activa PC amygdala DBS

INTERVENTIONS:
Device: Week 0 Medtronic 3387 electrodes/Activa PC amygdala DBS — Subjects undergo the placement of a Leksell (Elekta, Atlanta, GE) stereotactic frame. Electrode trajectory planned using stereotactic software (BrainLab, Germany). Traditional trans-frontal trajectory used to implant Medtronic #3387 DBS electrodes bilaterally in the BLn. A curvilinear incision will be made 3 cm lateral to midline and 1 cm in front of the coronal suture. A burr hole will be placed with a high-speed drill for placement of a Stimloc device to hold the electrode in place. The dura will be opened, coagulated back and the cortex exposed, coagulated, and pierced. The electrode will be introduced using a cannula. Each electrode contact will be stimulated up to 7 V to confirm the absence of immediate side effects; first left, then right. Electrode wires will be tunneled under skin to upper chest and connected to Medtronic Activa PC dual channel pulse generator. Both groups keep stimulators off until week 0, then this group has stimulators turned on.
  Other Names: Implanted Hardware (Medtronic, Minneapolis, MN); DBS electrodes 3387; Stimloc device to hold the electrode in place; Activa PC dual channel pulse generator
  Arms: Week 0 Medtronic 3387 electrodes/Activa PC amygdala DBS
Device: Week 12 Medtronic 3387 electrodes/Activa PC amygdala DBS — Subjects undergo the placement of a Leksell (Elekta, Atlanta, GE) stereotactic frame. Electrode trajectory planned using stereotactic software (BrainLab, Germany). Traditional trans-frontal trajectory used to implant Medtronic #3387 DBS electrodes bilaterally in the BLn. A curvilinear incision will be made 3 cm lateral to midline and 1 cm in front of the coronal suture. A burr hole will be placed with a high-speed drill for placement of a Stimloc device to hold the electrode in place. The dura will be opened, coagulated back and the cortex exposed, coagulated, and pierced. The electrode will be introduced using a cannula. Each electrode contact will be stimulated up to 7 V to confirm the absence of immediate side effects; first left, then right. Electrode wires will be tunneled under skin to upper chest and connected to Medtronic Activa PC dual channel pulse generator. Both groups keep stimulators off until week 0. This group has stimulators turned on at week 12.
  Other Names: Implanted Hardware (Medtronic, Minneapolis, MN); DBS electrodes 3387; Stimloc device to hold the electrode in place; Activa PC dual channel pulse generator

SUMMARY:
The purpose of this study is to determine whether deep brain stimulation of the basolateral nucleus (BLn) of the amygdala, on both sides of the brain, can safely reduce symptoms of post-traumatic stress disorder (PTSD) in combat veterans whose condition has not improved despite extensive treatment with currently available medication and psychotherapy interventions.

DETAILED DESCRIPTION:
For this pilot feasibility study, combat veterans whose PTSD has been associated with severe symptomatic suffering and functional impairment, despite treatment with all currently available pharmacological and psychotherapeutic treatments, will be recruited from clinics at a large, academically affiliated VA facility. An extensive screening over an extended baseline by the study psychiatrist and neurosurgeon will be conducted using standard interviews and clinical rating scales. Eligible subjects are required to have a cohabiting significant other willing to participate in safety and function monitoring throughout the study.

After successful completion of baseline eligibility requirements, comprehensive neuropsychological testing will be performed, as will structural MRI and FDG PET/CT of the amygdala, insula and medial Prefrontal cortex. PET/CT will be performed and analyzed by a nuclear medicine specialist collaborator familiar with this type of imaging research. Six consenting subjects meeting all eligibility criteria will then receive bilateral basolateral nucleus of the amygdala (BlnA) implantation of Medtronic Activa Primary Cell (PC) implantable deep brain stimulator systems (purchased through the VA Merit Review Grant) by functional neurosurgeons specialized in the procedure. This will be done during a 3-4 day inpatient stay on the VA Greater Los Angeles Neurosurgical Service. After a month of weekly safety monitoring with stimulators off, subjects will be will be hospitalized for 1 day on the Neurology Service's electroencephalography (EEG) telemetry unit, under the care and supervision of an epilepsy specialist neurologist who is a co-investigator in the study, for stimulator initiation. Stimulator settings will be adjusted by the study clinical neurophysiologist while patients are monitored by the study neurologist and psychiatrist. Only stimulator settings that do not cause epileptiform discharges, or potentially significant adverse psychiatric or medical (e.g., blood pressure, heart rate) changes will be used over the subsequent long-term follow-up.

After the EEG telemetry safety check, subjects will be randomized (3/3) to either have their stimulators turned on then (Week 0), or 3 months later (week 12). This staggered onset double-blind design has been used in other DBS trials in psychiatry. After week 0, for the next 2 years, subjects will be followed at regular intervals (weekly for 5 months, then monthly for 7 months, then quarterly for 12 months) by a psychiatrist, neurosurgeon, neurologist and neurophysiologist who will conduct an extensive battery of psychiatric and neurological testing (including periodic EEG recordings), as well as significant other interviews, while stimulator settings are adjusted based on standardized rating scale outcomes and adverse effects so as to optimize treatment outcome. The principal study hypothesis is that the symptomatic and functional benefits of chronic stimulation will outweigh the risks and adverse-effects, and that symptomatic improvement will be greater, without unacceptable adverse effects, in subjects with week 0, compared to week 12 stimulator initiation. Neuropsychological testing will be repeated after 6 months of stimulation to assess changes in cognitive function. Functional neuroimaging with PET/CT will be repeated after a year of stimulation to assess changes in the activity of brain regions known to function abnormally in PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 25-65 years.
* Able to give informed consent in accordance with institutional policies and participate in the 2-year follow-up, involving assessments and stimulator adjustments.
* Patients must be stable on their current psychotropic medication for a period of 2 months before implantation and agree to not increase dosages or add any new medications for the first 6 months of the study, unless medically necessary.
* Chart diagnosis of chronic and treatment-refractory PTSD as the principal psychiatric diagnosis and cause of distress and social/occupational impairment.
* Confirmation of PTSD as the primary psychiatric diagnosis by the study psychiatrist via clinical interview and CAPS.
* Confirmation of combat trauma exposure via military record review and a Combat Exposure Scale score > 9.
* Minimum 5 year total illness duration, with no 6 month period of clinical remission during the 5 years prior to entry in the study.
* Clinical record documentation of non-response to at least 2 of the following antidepressants, alone or in combination, at maximally tolerated FDA recommended doses for ≥ 6 months: sertraline, paroxetine, fluoxetine, citalopram, escitalopram, amitriptyline, imipramine, nortriptyline, desipramine, clomipramine, phenelzine, tranylcypromine, venlafaxine, mirtazapine. Antidepressant trials must include at least one SSRI and one SNRI or TCA at maximally tolerated FDA recommended doses for a minimum of 3 months.
* A minimum 3 month trial of prazosin at 10 mg per day or, if less, maximally tolerated FDA recommended doses, unless considered contraindicated based on co-morbid medical conditions or concomitant medications.
* Trial of at least 3 months of one of the following: lithium, divalproex sodium, carbamazepine, lamotrigine, olanzapine, risperidone, bupropion either alone or in conjunction with one or more of the agents in #8 and # 9 above.
* 6 months of continuous individual psychotherapy, conducted at least twice monthly for minimum 45 minute sessions, and consisting of a) clinician-defined cognitive-behavioural psychotherapy directed toward reducing conditioned fear symptoms of PTSD; b) cognitive processing psychotherapy for PTSD; c) prolonged exposure therapy for PTSD (imaginal, in vivo, and/or virtual reality); or d) Eye movement desensitization and reprocessing therapy for PTSD including a trauma exposure component, with chart documentation of inadequate benefit despite concerted effort. Other forms of individual or group psychotherapy are permitted but not required for inclusion. (Patients who are unable to complete 6 months of psychotherapy may be included if the cause of treatment cessation was that the risks of further treatment, including intense psychological suffering, outweighed the potential benefits of continuing the treatment).
* All evidence based psychotherapy for PTSD (cognitive behavioural, cognitive processing, prolonged exposure, eye movement desensitization) has been completed a minimum of 3 months prior to enrollment.
* Minimum baseline CAPS17 of 85 at entry, with a) scores of at least 4 (combined frequency and severity) on at least one symptom from each cluster (intrusion, avoidance and hyperarousal); b) score of 5 or more on CAPS17 items 4 or 5 (intense psychological distress or physiological reactivity on exposure to a reminder of the traumatic event); and c) no questionable validity (QV) rating greater than 1 on any CAPS item.
* Clinically significant impairment in occupational functioning due to PTSD, manifested by one or more of the following: a) Total federal (service connected ≥ 70%), or State (SSI) disability compensation for at least the past 2 years for PTSD; b) global assessment of functioning score ≤ 45; c) no period of full time gainful employment ≥ 3 months in the past 5 years.
* Clinically significant impairment in social functioning due to PTSD, manifested by one or more of the following: a) little or no social activity outside the household other than as necessary for medical appointments, practical matters such as grocery shopping, or to interact with other veterans; b) reliable description by a spouse or significant other, living with the patient, of repeated avoidance/refusal to participate in customary social engagements with friends, family or for recreational activities due to PTSD; c) two or more verbal or physical interpersonal altercations within the past year requiring another person's intervention to prevent further escalation, or involving law enforcement
* Cohabitation with a spouse or significant other adult person who a) can confirm the symptoms and impairment from PTSD and lack of significant symptomatic remission in the past 5 years; and b) is willing to participate with the study psychiatrist in answering questions for the life functioning in PTSD scale (LFIPS) at scheduled follow-up visits; and c) is willing to report unexpected adverse neurological or psychiatric events to study investigators and if advised by study investigators, assist the patient in accessing necessary services to address these.
* Willingness to have unexpected neurological or psychiatric symptom shared with the study psychiatrists and other study clinicians.
* Other medical conditions must be stable for at least 1 year, (conditions that require intermittent use of steroids or chemotherapy are excluded).

Exclusion Criteria:

* Suicide attempt in the last 2 years and/or presence of a suicide plan (an answer of "Yes" to Question C4 in Section C-Suicidality of MINI International Neuropsychiatric Interview);
* Psychosis or bipolar disorder; significant acute or ongoing risk for violence;
* Patients primarily diagnosed with DSM-IV-TR Axis I disorder other than PTSD as determined by the MINI;
* Within the 3 months prior to enrollment, subject has started a new psychotherapy program;
* Alcohol or illicit substance use disorder within the last 6 months, unstable remission of substance abuse, or chart evidence that co-morbid substance use disorder could account for lack of treatment response;
* Current significant neurological conditions, including epilepsy, stroke, movement disorder; history of serious head injury with loss of consciousness
* Uncontrolled medical condition including cardiovascular problems and diabetes;
* Uncontrolled chronic pain;
* Baseline Montgomery Asberg Depression Rating Scale (MADRS) of ≥ 28;
* Use of warfarin;
* Significant abnormality on preoperative structural brain MRI;
* ECT in the past 6 months;
* Contraindications to MRIs or the need for recurrent body MRIs;
* Immunosuppression;
* High risk for surgery;
* Current pursuit of new or increased disability compensation for PTSD;
* Has cardiac pacemaker/defibrillator, implanted medication pump, intra-cardiac lines, any intracranial implants (aneurysm clip, shunt, cochlear implant, electrodes) or other implanted stimulator;
* Patient has had past cranial neurosurgery;
* Patient unable to discontinue therapeutic diathermy;
* Use of other investigational drugs or psychotropic herbs within 30 days of baseline.

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The Clinician-Administered PTSD scale (CAPS) will be the primary outcome measure. A clinical response will be defined as a reduction of 30 % in CAPSSx from baseline to 12 months post-stimulation, without adverse events leading to stopping stimulation. | 12 months
  This is a standardized structured, clinician administered interview that includes both questions confirming the diagnosis of PTSD (CAPSDx) as well as symptom severity over specified time periods (lifetime, past week or past month) based on the 17 symptoms of PTSD in DSM-III/II-R and IV across clusters of recurrence, avoidance/numbing and hyper-arousal symptoms (CAPS1-17 or CAPSSx).

SECONDARY OUTCOMES:
The Clinician-Administered PTSD scale (CAPS) change from week 0 | 1 month
  This is a standardized structured, clinician administered interview that includes both questions confirming the diagnosis of PTSD (CAPSDx) as well as symptom severity over specified time periods (lifetime, past week or past month) based on the 17 symptoms of PTSD in DSM-III/II-R and IV across clusters of recurrence, avoidance/numbing and hyper-arousal symptoms (CAPS1-17 or CAPSSx).
The Clinician-Administered PTSD scale (CAPS) change from week 0 | 2months
  This is a standardized structured, clinician administered interview that includes both questions confirming the diagnosis of PTSD (CAPSDx) as well as symptom severity over specified time periods (lifetime, past week or past month) based on the 17 symptoms of PTSD in DSM-III/II-R and IV across clusters of recurrence, avoidance/numbing and hyper-arousal symptoms (CAPS1-17 or CAPSSx).
The Clinician-Administered PTSD scale (CAPS) change from week 0 | 3 months
  This is a standardized structured, clinician administered interview that includes both questions confirming the diagnosis of PTSD (CAPSDx) as well as symptom severity over specified time periods (lifetime, past week or past month) based on the 17 symptoms of PTSD in DSM-III/II-R and IV across clusters of recurrence, avoidance/numbing and hyper-arousal symptoms (CAPS1-17 or CAPSSx).
The Clinician-Administered PTSD scale (CAPS) change from week 0 | 4 months
  This is a standardized structured, clinician administered interview that includes both questions confirming the diagnosis of PTSD (CAPSDx) as well as symptom severity over specified time periods (lifetime, past week or past month) based on the 17 symptoms of PTSD in DSM-III/II-R and IV across clusters of recurrence, avoidance/numbing and hyper-arousal symptoms (CAPS1-17 or CAPSSx).
The Clinician-Administered PTSD scale (CAPS) change from week 0 | 5 months
  This is a standardized structured, clinician administered interview that includes both questions confirming the diagnosis of PTSD (CAPSDx) as well as symptom severity over specified time periods (lifetime, past week or past month) based on the 17 symptoms of PTSD in DSM-III/II-R and IV across clusters of recurrence, avoidance/numbing and hyper-arousal symptoms (CAPS1-17 or CAPSSx).
The Clinician-Administered PTSD scale (CAPS) change from week 0 | 6 months
  This is a standardized structured, clinician administered interview that includes both questions confirming the diagnosis of PTSD (CAPSDx) as well as symptom severity over specified time periods (lifetime, past week or past month) based on the 17 symptoms of PTSD in DSM-III/II-R and IV across clusters of recurrence, avoidance/numbing and hyper-arousal symptoms (CAPS1-17 or CAPSSx).
The Clinician-Administered PTSD scale (CAPS) change from week 0 | 7 months
  This is a standardized structured, clinician administered interview that includes both questions confirming the diagnosis of PTSD (CAPSDx) as well as symptom severity over specified time periods (lifetime, past week or past month) based on the 17 symptoms of PTSD in DSM-III/II-R and IV across clusters of recurrence, avoidance/numbing and hyper-arousal symptoms (CAPS1-17 or CAPSSx).
The Clinician-Administered PTSD scale (CAPS) change from week 0 | 8 months
  This is a standardized structured, clinician administered interview that includes both questions confirming the diagnosis of PTSD (CAPSDx) as well as symptom severity over specified time periods (lifetime, past week or past month) based on the 17 symptoms of PTSD in DSM-III/II-R and IV across clusters of recurrence, avoidance/numbing and hyper-arousal symptoms (CAPS1-17 or CAPSSx).
The Clinician-Administered PTSD scale (CAPS) change from week 0 | 9 months
  This is a standardized structured, clinician administered interview that includes both questions confirming the diagnosis of PTSD (CAPSDx) as well as symptom severity over specified time periods (lifetime, past week or past month) based on the 17 symptoms of PTSD in DSM-III/II-R and IV across clusters of recurrence, avoidance/numbing and hyper-arousal symptoms (CAPS1-17 or CAPSSx).
The Clinician-Administered PTSD scale (CAPS) change from week 0 | 10 months
  This is a standardized structured, clinician administered interview that includes both questions confirming the diagnosis of PTSD (CAPSDx) as well as symptom severity over specified time periods (lifetime, past week or past month) based on the 17 symptoms of PTSD in DSM-III/II-R and IV across clusters of recurrence, avoidance/numbing and hyper-arousal symptoms (CAPS1-17 or CAPSSx).
The Clinician-Administered PTSD scale (CAPS) change from week 0 | 11 months
  This is a standardized structured, clinician administered interview that includes both questions confirming the diagnosis of PTSD (CAPSDx) as well as symptom severity over specified time periods (lifetime, past week or past month) based on the 17 symptoms of PTSD in DSM-III/II-R and IV across clusters of recurrence, avoidance/numbing and hyper-arousal symptoms (CAPS1-17 or CAPSSx).
The Clinician-Administered PTSD scale (CAPS) change from week 0 | 13 months
  This is a standardized structured, clinician administered interview that includes both questions confirming the diagnosis of PTSD (CAPSDx) as well as symptom severity over specified time periods (lifetime, past week or past month) based on the 17 symptoms of PTSD in DSM-III/II-R and IV across clusters of recurrence, avoidance/numbing and hyper-arousal symptoms (CAPS1-17 or CAPSSx).
The Clinician-Administered PTSD scale (CAPS) change from week 0 | 14 months
  This is a standardized structured, clinician administered interview that includes both questions confirming the diagnosis of PTSD (CAPSDx) as well as symptom severity over specified time periods (lifetime, past week or past month) based on the 17 symptoms of PTSD in DSM-III/II-R and IV across clusters of recurrence, avoidance/numbing and hyper-arousal symptoms (CAPS1-17 or CAPSSx).
The Clinician-Administered PTSD scale (CAPS) change from week 0 | 15 months
  This is a standardized structured, clinician administered interview that includes both questions confirming the diagnosis of PTSD (CAPSDx) as well as symptom severity over specified time periods (lifetime, past week or past month) based on the 17 symptoms of PTSD in DSM-III/II-R and IV across clusters of recurrence, avoidance/numbing and hyper-arousal symptoms (CAPS1-17 or CAPSSx).
The Clinician-Administered PTSD scale (CAPS) change from week 0 | 18 months
  This is a standardized structured, clinician administered interview that includes both questions confirming the diagnosis of PTSD (CAPSDx) as well as symptom severity over specified time periods (lifetime, past week or past month) based on the 17 symptoms of PTSD in DSM-III/II-R and IV across clusters of recurrence, avoidance/numbing and hyper-arousal symptoms (CAPS1-17 or CAPSSx).
The Clinician-Administered PTSD scale (CAPS) change from week 0 | 21 months
  This is a standardized structured, clinician administered interview that includes both questions confirming the diagnosis of PTSD (CAPSDx) as well as symptom severity over specified time periods (lifetime, past week or past month) based on the 17 symptoms of PTSD in DSM-III/II-R and IV across clusters of recurrence, avoidance/numbing and hyper-arousal symptoms (CAPS1-17 or CAPSSx).
The Clinician-Administered PTSD scale (CAPS) change from week 0 | 24 months
  This is a standardized structured, clinician administered interview that includes both questions confirming the diagnosis of PTSD (CAPSDx) as well as symptom severity over specified time periods (lifetime, past week or past month) based on the 17 symptoms of PTSD in DSM-III/II-R and IV across clusters of recurrence, avoidance/numbing and hyper-arousal symptoms (CAPS1-17 or CAPSSx).
Hamilton Anxiety Rating Scale (HAM-A) change from week 0 | 3 months
  Clinician administered scale to rate cross-sectional severity of generalized anxiety symptoms
Hamilton Anxiety Rating Scale (HAM-A) change from week 0 | 6 months
  Clinician administered scale to rate cross-sectional severity of generalized anxiety symptoms
Hamilton Anxiety Rating Scale (HAM-A) change from week 0 | 9 months
  Clinician administered scale to rate cross-sectional severity of generalized anxiety symptoms
Hamilton Anxiety Rating Scale (HAM-A) change from week 0 | 12 months
  Clinician administered scale to rate cross-sectional severity of generalized anxiety symptoms
Hamilton Anxiety Rating Scale (HAM-A) change from week 0 | 15 months
  Clinician administered scale to rate cross-sectional severity of generalized anxiety symptoms
Hamilton Anxiety Rating Scale (HAM-A) change from week 0 | 18 months
  Clinician administered scale to rate cross-sectional severity of generalized anxiety symptoms
Hamilton Anxiety Rating Scale (HAM-A) change from week 0 | 21 months
  Clinician administered scale to rate cross-sectional severity of generalized anxiety symptoms
Hamilton Anxiety Rating Scale (HAM-A) change from week 0 | 24 months
  Clinician administered scale to rate cross-sectional severity of generalized anxiety symptoms
Montgomery Asberg Depression Rating Scale (MADRS) change from week 0 | 1 month
  The MADRS is a 10 item clinician administered rating instrument with each item rated on a 7 point (0-6) scale to evaluate the severity of depressive symptoms in patients diagnosed with a depressive disorder. It is designed to evaluate for change in depressive state during treatment. Total scores range from 0-52 with score interpretation of: 7 recovered, 15 mild depression, 25 moderate depression, 31 severe and 44 very severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) change from week 0 | 3 months
  The MADRS is a 10 item clinician administered rating instrument with each item rated on a 7 point (0-6) scale to evaluate the severity of depressive symptoms in patients diagnosed with a depressive disorder. It is designed to evaluate for change in depressive state during treatment. Total scores range from 0-52 with score interpretation of: 7 recovered, 15 mild depression, 25 moderate depression, 31 severe and 44 very severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) change from week 0 | 4 months
  The MADRS is a 10 item clinician administered rating instrument with each item rated on a 7 point (0-6) scale to evaluate the severity of depressive symptoms in patients diagnosed with a depressive disorder. It is designed to evaluate for change in depressive state during treatment. Total scores range from 0-52 with score interpretation of: 7 recovered, 15 mild depression, 25 moderate depression, 31 severe and 44 very severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) change from week 0 | 5 months
  The MADRS is a 10 item clinician administered rating instrument with each item rated on a 7 point (0-6) scale to evaluate the severity of depressive symptoms in patients diagnosed with a depressive disorder. It is designed to evaluate for change in depressive state during treatment. Total scores range from 0-52 with score interpretation of: 7 recovered, 15 mild depression, 25 moderate depression, 31 severe and 44 very severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) change from week 0 | 6 months
  The MADRS is a 10 item clinician administered rating instrument with each item rated on a 7 point (0-6) scale to evaluate the severity of depressive symptoms in patients diagnosed with a depressive disorder. It is designed to evaluate for change in depressive state during treatment. Total scores range from 0-52 with score interpretation of: 7 recovered, 15 mild depression, 25 moderate depression, 31 severe and 44 very severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) change from week 0 | 7 months
  The MADRS is a 10 item clinician administered rating instrument with each item rated on a 7 point (0-6) scale to evaluate the severity of depressive symptoms in patients diagnosed with a depressive disorder. It is designed to evaluate for change in depressive state during treatment. Total scores range from 0-52 with score interpretation of: 7 recovered, 15 mild depression, 25 moderate depression, 31 severe and 44 very severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) change from week 0 | 8 months
  The MADRS is a 10 item clinician administered rating instrument with each item rated on a 7 point (0-6) scale to evaluate the severity of depressive symptoms in patients diagnosed with a depressive disorder. It is designed to evaluate for change in depressive state during treatment. Total scores range from 0-52 with score interpretation of: 7 recovered, 15 mild depression, 25 moderate depression, 31 severe and 44 very severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) change from week 0 | 9 months
  The MADRS is a 10 item clinician administered rating instrument with each item rated on a 7 point (0-6) scale to evaluate the severity of depressive symptoms in patients diagnosed with a depressive disorder. It is designed to evaluate for change in depressive state during treatment. Total scores range from 0-52 with score interpretation of: 7 recovered, 15 mild depression, 25 moderate depression, 31 severe and 44 very severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) change from week 0 | 10 months
  The MADRS is a 10 item clinician administered rating instrument with each item rated on a 7 point (0-6) scale to evaluate the severity of depressive symptoms in patients diagnosed with a depressive disorder. It is designed to evaluate for change in depressive state during treatment. Total scores range from 0-52 with score interpretation of: 7 recovered, 15 mild depression, 25 moderate depression, 31 severe and 44 very severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) change from week 0 | 11 months
  The MADRS is a 10 item clinician administered rating instrument with each item rated on a 7 point (0-6) scale to evaluate the severity of depressive symptoms in patients diagnosed with a depressive disorder. It is designed to evaluate for change in depressive state during treatment. Total scores range from 0-52 with score interpretation of: 7 recovered, 15 mild depression, 25 moderate depression, 31 severe and 44 very severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) change from week 0 | 12 months
  The MADRS is a 10 item clinician administered rating instrument with each item rated on a 7 point (0-6) scale to evaluate the severity of depressive symptoms in patients diagnosed with a depressive disorder. It is designed to evaluate for change in depressive state during treatment. Total scores range from 0-52 with score interpretation of: 7 recovered, 15 mild depression, 25 moderate depression, 31 severe and 44 very severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) change from week 0 | 13 months
  The MADRS is a 10 item clinician administered rating instrument with each item rated on a 7 point (0-6) scale to evaluate the severity of depressive symptoms in patients diagnosed with a depressive disorder. It is designed to evaluate for change in depressive state during treatment. Total scores range from 0-52 with score interpretation of: 7 recovered, 15 mild depression, 25 moderate depression, 31 severe and 44 very severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) change from week 0 | 14 months
  The MADRS is a 10 item clinician administered rating instrument with each item rated on a 7 point (0-6) scale to evaluate the severity of depressive symptoms in patients diagnosed with a depressive disorder. It is designed to evaluate for change in depressive state during treatment. Total scores range from 0-52 with score interpretation of: 7 recovered, 15 mild depression, 25 moderate depression, 31 severe and 44 very severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) change from week 0 | 15 months
  The MADRS is a 10 item clinician administered rating instrument with each item rated on a 7 point (0-6) scale to evaluate the severity of depressive symptoms in patients diagnosed with a depressive disorder. It is designed to evaluate for change in depressive state during treatment. Total scores range from 0-52 with score interpretation of: 7 recovered, 15 mild depression, 25 moderate depression, 31 severe and 44 very severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) change from week 0 | 18 months
  The MADRS is a 10 item clinician administered rating instrument with each item rated on a 7 point (0-6) scale to evaluate the severity of depressive symptoms in patients diagnosed with a depressive disorder. It is designed to evaluate for change in depressive state during treatment. Total scores range from 0-52 with score interpretation of: 7 recovered, 15 mild depression, 25 moderate depression, 31 severe and 44 very severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) change from week 0 | 21 months
  The MADRS is a 10 item clinician administered rating instrument with each item rated on a 7 point (0-6) scale to evaluate the severity of depressive symptoms in patients diagnosed with a depressive disorder. It is designed to evaluate for change in depressive state during treatment. Total scores range from 0-52 with score interpretation of: 7 recovered, 15 mild depression, 25 moderate depression, 31 severe and 44 very severe depression.
Montgomery Asberg Depression Rating Scale (MADRS) change from week 0 | 24 months
  The MADRS is a 10 item clinician administered rating instrument with each item rated on a 7 point (0-6) scale to evaluate the severity of depressive symptoms in patients diagnosed with a depressive disorder. It is designed to evaluate for change in depressive state during treatment. Total scores range from 0-52 with score interpretation of: 7 recovered, 15 mild depression, 25 moderate depression, 31 severe and 44 very severe depression.
Young Mania Rating Scale (YMRS) change from week 0 | 1 month
  The YMRS is an 11-item clinician-administered cross-sectional rating instrument used to assess the severity of mania in patients with a diagnosis of bipolar disorder. The 11 items are: Elevated Mood, Increased Motor Activity/Energy, Sexual Interest, Sleep, Irritability, Speech (Rate and Amount), Language - Thought Disorder, Content, Disruptive/Aggressive Behaviour, Appearance and Insight.
  Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score).
Young Mania Rating Scale (YMRS) change from week 0 | 2 months
  The YMRS is an 11-item clinician-administered cross-sectional rating instrument used to assess the severity of mania in patients with a diagnosis of bipolar disorder. The 11 items are: Elevated Mood, Increased Motor Activity/Energy, Sexual Interest, Sleep, Irritability, Speech (Rate and Amount), Language - Thought Disorder, Content, Disruptive/Aggressive Behaviour, Appearance and Insight.
  Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score).
Young Mania Rating Scale (YMRS) change from week 0 | 3 months
  The YMRS is an 11-item clinician-administered cross-sectional rating instrument used to assess the severity of mania in patients with a diagnosis of bipolar disorder. The 11 items are: Elevated Mood, Increased Motor Activity/Energy, Sexual Interest, Sleep, Irritability, Speech (Rate and Amount), Language - Thought Disorder, Content, Disruptive/Aggressive Behaviour, Appearance and Insight.
  Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score).
Young Mania Rating Scale (YMRS) change from week 0 | 4 months
  The YMRS is an 11-item clinician-administered cross-sectional rating instrument used to assess the severity of mania in patients with a diagnosis of bipolar disorder. The 11 items are: Elevated Mood, Increased Motor Activity/Energy, Sexual Interest, Sleep, Irritability, Speech (Rate and Amount), Language - Thought Disorder, Content, Disruptive/Aggressive Behaviour, Appearance and Insight.
  Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score).
Young Mania Rating Scale (YMRS) change from week 0 | 5 months
  The YMRS is an 11-item clinician-administered cross-sectional rating instrument used to assess the severity of mania in patients with a diagnosis of bipolar disorder. The 11 items are: Elevated Mood, Increased Motor Activity/Energy, Sexual Interest, Sleep, Irritability, Speech (Rate and Amount), Language - Thought Disorder, Content, Disruptive/Aggressive Behaviour, Appearance and Insight.
  Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score).
Young Mania Rating Scale (YMRS) change from week 0 | 6 months
  The YMRS is an 11-item clinician-administered cross-sectional rating instrument used to assess the severity of mania in patients with a diagnosis of bipolar disorder. The 11 items are: Elevated Mood, Increased Motor Activity/Energy, Sexual Interest, Sleep, Irritability, Speech (Rate and Amount), Language - Thought Disorder, Content, Disruptive/Aggressive Behaviour, Appearance and Insight.
  Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score).
Young Mania Rating Scale (YMRS) change from week 0 | 7 months
  The YMRS is an 11-item clinician-administered cross-sectional rating instrument used to assess the severity of mania in patients with a diagnosis of bipolar disorder. The 11 items are: Elevated Mood, Increased Motor Activity/Energy, Sexual Interest, Sleep, Irritability, Speech (Rate and Amount), Language - Thought Disorder, Content, Disruptive/Aggressive Behaviour, Appearance and Insight.
  Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score).
Young Mania Rating Scale (YMRS) change from week 0 | 8 months
  The YMRS is an 11-item clinician-administered cross-sectional rating instrument used to assess the severity of mania in patients with a diagnosis of bipolar disorder. The 11 items are: Elevated Mood, Increased Motor Activity/Energy, Sexual Interest, Sleep, Irritability, Speech (Rate and Amount), Language - Thought Disorder, Content, Disruptive/Aggressive Behaviour, Appearance and Insight.
  Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score).
Young Mania Rating Scale (YMRS) change from week 0 | 9 months
  The YMRS is an 11-item clinician-administered cross-sectional rating instrument used to assess the severity of mania in patients with a diagnosis of bipolar disorder. The 11 items are: Elevated Mood, Increased Motor Activity/Energy, Sexual Interest, Sleep, Irritability, Speech (Rate and Amount), Language - Thought Disorder, Content, Disruptive/Aggressive Behaviour, Appearance and Insight.
  Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score).
Young Mania Rating Scale (YMRS) change from week 0 | 10 months
  The YMRS is an 11-item clinician-administered cross-sectional rating instrument used to assess the severity of mania in patients with a diagnosis of bipolar disorder. The 11 items are: Elevated Mood, Increased Motor Activity/Energy, Sexual Interest, Sleep, Irritability, Speech (Rate and Amount), Language - Thought Disorder, Content, Disruptive/Aggressive Behaviour, Appearance and Insight.
  Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score).
Young Mania Rating Scale (YMRS) change from week 0 | 11 months
  The YMRS is an 11-item clinician-administered cross-sectional rating instrument used to assess the severity of mania in patients with a diagnosis of bipolar disorder. The 11 items are: Elevated Mood, Increased Motor Activity/Energy, Sexual Interest, Sleep, Irritability, Speech (Rate and Amount), Language - Thought Disorder, Content, Disruptive/Aggressive Behaviour, Appearance and Insight.
  Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score).
Young Mania Rating Scale (YMRS) change from week 0 | 12 months
  The YMRS is an 11-item clinician-administered cross-sectional rating instrument used to assess the severity of mania in patients with a diagnosis of bipolar disorder. The 11 items are: Elevated Mood, Increased Motor Activity/Energy, Sexual Interest, Sleep, Irritability, Speech (Rate and Amount), Language - Thought Disorder, Content, Disruptive/Aggressive Behaviour, Appearance and Insight.
  Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score).
Young Mania Rating Scale (YMRS) change from week 0 | 13 months
  The YMRS is an 11-item clinician-administered cross-sectional rating instrument used to assess the severity of mania in patients with a diagnosis of bipolar disorder. The 11 items are: Elevated Mood, Increased Motor Activity/Energy, Sexual Interest, Sleep, Irritability, Speech (Rate and Amount), Language - Thought Disorder, Content, Disruptive/Aggressive Behaviour, Appearance and Insight.
  Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score).
Young Mania Rating Scale (YMRS) change from week 0 | 14 months
  The YMRS is an 11-item clinician-administered cross-sectional rating instrument used to assess the severity of mania in patients with a diagnosis of bipolar disorder. The 11 items are: Elevated Mood, Increased Motor Activity/Energy, Sexual Interest, Sleep, Irritability, Speech (Rate and Amount), Language - Thought Disorder, Content, Disruptive/Aggressive Behaviour, Appearance and Insight.
  Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score).
Young Mania Rating Scale (YMRS) change from week 0 | 15 months
  The YMRS is an 11-item clinician-administered cross-sectional rating instrument used to assess the severity of mania in patients with a diagnosis of bipolar disorder. The 11 items are: Elevated Mood, Increased Motor Activity/Energy, Sexual Interest, Sleep, Irritability, Speech (Rate and Amount), Language - Thought Disorder, Content, Disruptive/Aggressive Behaviour, Appearance and Insight.
  Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score).
Young Mania Rating Scale (YMRS) change from week 0 | 18 months
  The YMRS is an 11-item clinician-administered cross-sectional rating instrument used to assess the severity of mania in patients with a diagnosis of bipolar disorder. The 11 items are: Elevated Mood, Increased Motor Activity/Energy, Sexual Interest, Sleep, Irritability, Speech (Rate and Amount), Language - Thought Disorder, Content, Disruptive/Aggressive Behaviour, Appearance and Insight.
  Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score).
Young Mania Rating Scale (YMRS) change from week 0 | 21 months
  The YMRS is an 11-item clinician-administered cross-sectional rating instrument used to assess the severity of mania in patients with a diagnosis of bipolar disorder. The 11 items are: Elevated Mood, Increased Motor Activity/Energy, Sexual Interest, Sleep, Irritability, Speech (Rate and Amount), Language - Thought Disorder, Content, Disruptive/Aggressive Behaviour, Appearance and Insight.
  Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score).
Young Mania Rating Scale (YMRS) change from week 0 | 24 months
  The YMRS is an 11-item clinician-administered cross-sectional rating instrument used to assess the severity of mania in patients with a diagnosis of bipolar disorder. The 11 items are: Elevated Mood, Increased Motor Activity/Energy, Sexual Interest, Sleep, Irritability, Speech (Rate and Amount), Language - Thought Disorder, Content, Disruptive/Aggressive Behaviour, Appearance and Insight.
  Ratings are based on patient self-reporting, combined with clinician observation (accorded greater score).
Columbia-Suicide Severity Rating Scale (C-SSRS) change from week 0 | 1 month
  The C-SSRS is a semi-structured clinical interview that utilizes a set of prompts and questions to help an interviewer assess the full range of suicidal ideation and behavior, and the intensity of ideation, which helps an interviewer get more complete information on suicide risk.
Columbia-Suicide Severity Rating Scale (C-SSRS) change from week 0 | 2 months
  The C-SSRS is a semi-structured clinical interview that utilizes a set of prompts and questions to help an interviewer assess the full range of suicidal ideation and behavior, and the intensity of ideation, which helps an interviewer get more complete information on suicide risk.
Columbia-Suicide Severity Rating Scale (C-SSRS) change from week 0 | 3 months
  The C-SSRS is a semi-structured clinical interview that utilizes a set of prompts and questions to help an interviewer assess the full range of suicidal ideation and behavior, and the intensity of ideation, which helps an interviewer get more complete information on suicide risk.
Columbia-Suicide Severity Rating Scale (C-SSRS) change from week 0 | 4 months
  The C-SSRS is a semi-structured clinical interview that utilizes a set of prompts and questions to help an interviewer assess the full range of suicidal ideation and behavior, and the intensity of ideation, which helps an interviewer get more complete information on suicide risk.
Columbia-Suicide Severity Rating Scale (C-SSRS) change from week 0 | 5 months
  The C-SSRS is a semi-structured clinical interview that utilizes a set of prompts and questions to help an interviewer assess the full range of suicidal ideation and behavior, and the intensity of ideation, which helps an interviewer get more complete information on suicide risk.
Columbia-Suicide Severity Rating Scale (C-SSRS) change from week 0 | 6 months
  The C-SSRS is a semi-structured clinical interview that utilizes a set of prompts and questions to help an interviewer assess the full range of suicidal ideation and behavior, and the intensity of ideation, which helps an interviewer get more complete information on suicide risk.
Columbia-Suicide Severity Rating Scale (C-SSRS) change from week 0 | 9 months
  The C-SSRS is a semi-structured clinical interview that utilizes a set of prompts and questions to help an interviewer assess the full range of suicidal ideation and behavior, and the intensity of ideation, which helps an interviewer get more complete information on suicide risk.
Columbia-Suicide Severity Rating Scale (C-SSRS) change from week 0 | 12 months
  The C-SSRS is a semi-structured clinical interview that utilizes a set of prompts and questions to help an interviewer assess the full range of suicidal ideation and behavior, and the intensity of ideation, which helps an interviewer get more complete information on suicide risk.
Columbia-Suicide Severity Rating Scale (C-SSRS) change from week 0 | 15 months
  The C-SSRS is a semi-structured clinical interview that utilizes a set of prompts and questions to help an interviewer assess the full range of suicidal ideation and behavior, and the intensity of ideation, which helps an interviewer get more complete information on suicide risk.
Columbia-Suicide Severity Rating Scale (C-SSRS) change from week 0 | 18 months
  The C-SSRS is a semi-structured clinical interview that utilizes a set of prompts and questions to help an interviewer assess the full range of suicidal ideation and behavior, and the intensity of ideation, which helps an interviewer get more complete information on suicide risk.
Columbia-Suicide Severity Rating Scale (C-SSRS) change from week 0 | 21 months
  The C-SSRS is a semi-structured clinical interview that utilizes a set of prompts and questions to help an interviewer assess the full range of suicidal ideation and behavior, and the intensity of ideation, which helps an interviewer get more complete information on suicide risk.
Columbia-Suicide Severity Rating Scale (C-SSRS) change from week 0 | 24 months
  The C-SSRS is a semi-structured clinical interview that utilizes a set of prompts and questions to help an interviewer assess the full range of suicidal ideation and behavior, and the intensity of ideation, which helps an interviewer get more complete information on suicide risk.
Clinical Global Impression and Improvement Scales (CGI-S and CGI-I) change from week 0 | 1 month
  Standardized clinician-administered, cross-sectional assessment of global severity (CGI-S) of PTSD symptomatic status and improvement (CGI-I) from baseline on ordinal 7 point scale.
Clinical Global Impression and Improvement Scales (CGI-S and CGI-I) change from week 0 | 2 months
  Standardized clinician-administered, cross-sectional assessment of global severity (CGI-S) of PTSD symptomatic status and improvement (CGI-I) from baseline on ordinal 7 point scale.
Clinical Global Impression and Improvement Scales (CGI-S and CGI-I) change from week 0 | 3 months
  Standardized clinician-administered, cross-sectional assessment of global severity (CGI-S) of PTSD symptomatic status and improvement (CGI-I) from baseline on ordinal 7 point scale.
Clinical Global Impression and Improvement Scales (CGI-S and CGI-I) change from week 0 | 4 months
  Standardized clinician-administered, cross-sectional assessment of global severity (CGI-S) of PTSD symptomatic status and improvement (CGI-I) from baseline on ordinal 7 point scale.
Clinical Global Impression and Improvement Scales (CGI-S and CGI-I) change from week 0 | 5 months
  Standardized clinician-administered, cross-sectional assessment of global severity (CGI-S) of PTSD symptomatic status and improvement (CGI-I) from baseline on ordinal 7 point scale.
Clinical Global Impression and Improvement Scales (CGI-S and CGI-I) change from week 0 | 6 months
  Standardized clinician-administered, cross-sectional assessment of global severity (CGI-S) of PTSD symptomatic status and improvement (CGI-I) from baseline on ordinal 7 point scale.
Clinical Global Impression and Improvement Scales (CGI-S and CGI-I) change from week 0 | 7 months
  Standardized clinician-administered, cross-sectional assessment of global severity (CGI-S) of PTSD symptomatic status and improvement (CGI-I) from baseline on ordinal 7 point scale.
Clinical Global Impression and Improvement Scales (CGI-S and CGI-I) change from week 0 | 8 months
  Standardized clinician-administered, cross-sectional assessment of global severity (CGI-S) of PTSD symptomatic status and improvement (CGI-I) from baseline on ordinal 7 point scale.
Clinical Global Impression and Improvement Scales (CGI-S and CGI-I) change from week 0 | 9 months
  Standardized clinician-administered, cross-sectional assessment of global severity (CGI-S) of PTSD symptomatic status and improvement (CGI-I) from baseline on ordinal 7 point scale.
Clinical Global Impression and Improvement Scales (CGI-S and CGI-I) change from week 0 | 11 months
  Standardized clinician-administered, cross-sectional assessment of global severity (CGI-S) of PTSD symptomatic status and improvement (CGI-I) from baseline on ordinal 7 point scale.
Clinical Global Impression and Improvement Scales (CGI-S and CGI-I) change from week 0 | 12 months
  Standardized clinician-administered, cross-sectional assessment of global severity (CGI-S) of PTSD symptomatic status and improvement (CGI-I) from baseline on ordinal 7 point scale.
Clinical Global Impression and Improvement Scales (CGI-S and CGI-I) change from week 0 | 13 months
  Standardized clinician-administered, cross-sectional assessment of global severity (CGI-S) of PTSD symptomatic status and improvement (CGI-I) from baseline on ordinal 7 point scale.
Clinical Global Impression and Improvement Scales (CGI-S and CGI-I) change from week 0 | 14 months
  Standardized clinician-administered, cross-sectional assessment of global severity (CGI-S) of PTSD symptomatic status and improvement (CGI-I) from baseline on ordinal 7 point scale.
Clinical Global Impression and Improvement Scales (CGI-S and CGI-I) change from week 0 | 15 months
  Standardized clinician-administered, cross-sectional assessment of global severity (CGI-S) of PTSD symptomatic status and improvement (CGI-I) from baseline on ordinal 7 point scale.
Clinical Global Impression and Improvement Scales (CGI-S and CGI-I) change from week 0 | 18 months
  Standardized clinician-administered, cross-sectional assessment of global severity (CGI-S) of PTSD symptomatic status and improvement (CGI-I) from baseline on ordinal 7 point scale.
Clinical Global Impression and Improvement Scales (CGI-S and CGI-I) change from week 0 | 21 months
  Standardized clinician-administered, cross-sectional assessment of global severity (CGI-S) of PTSD symptomatic status and improvement (CGI-I) from baseline on ordinal 7 point scale.
Clinical Global Impression and Improvement Scales (CGI-S and CGI-I) change from week 0 | 24 months
  Standardized clinician-administered, cross-sectional assessment of global severity (CGI-S) of PTSD symptomatic status and improvement (CGI-I) from baseline on ordinal 7 point scale.
Veterans Quality of Life Assessment Scale (SF-36v) change from week 0 | 3 months
  Standardized, patient-rated cross-sectional scale measuring subjective physical and emotional health across 8 domains: general health (GH), physical function (PF), role limitations due to physical health (RP), bodily pain (BP), mental health (MH), role limitations due to emotional problems (RE), energy/vitality (VT), and social functioning (SF). The RP and RE scales have been modified in the veterans version from yes/no responses to five point ordinal choices. Otherwise the scale is comparable to the Medical Outcomes SF-36 functional assessment scale.
Veterans Quality of Life Assessment Scale (SF-36v) change from week 0 | 6 months
  Standardized, patient-rated cross-sectional scale measuring subjective physical and emotional health across 8 domains: general health (GH), physical function (PF), role limitations due to physical health (RP), bodily pain (BP), mental health (MH), role limitations due to emotional problems (RE), energy/vitality (VT), and social functioning (SF). The RP and RE scales have been modified in the veterans version from yes/no responses to five point ordinal choices. Otherwise the scale is comparable to the Medical Outcomes SF-36 functional assessment scale.
Veterans Quality of Life Assessment Scale (SF-36v) change from week 0 | 9 months
  Standardized, patient-rated cross-sectional scale measuring subjective physical and emotional health across 8 domains: general health (GH), physical function (PF), role limitations due to physical health (RP), bodily pain (BP), mental health (MH), role limitations due to emotional problems (RE), energy/vitality (VT), and social functioning (SF). The RP and RE scales have been modified in the veterans version from yes/no responses to five point ordinal choices. Otherwise the scale is comparable to the Medical Outcomes SF-36 functional assessment scale.
Veterans Quality of Life Assessment Scale (SF-36v) change from week 0 | 12 months
  Standardized, patient-rated cross-sectional scale measuring subjective physical and emotional health across 8 domains: general health (GH), physical function (PF), role limitations due to physical health (RP), bodily pain (BP), mental health (MH), role limitations due to emotional problems (RE), energy/vitality (VT), and social functioning (SF). The RP and RE scales have been modified in the veterans version from yes/no responses to five point ordinal choices. Otherwise the scale is comparable to the Medical Outcomes SF-36 functional assessment scale.
Veterans Quality of Life Assessment Scale (SF-36v) change from week 0 | 15 months
  Standardized, patient-rated cross-sectional scale measuring subjective physical and emotional health across 8 domains: general health (GH), physical function (PF), role limitations due to physical health (RP), bodily pain (BP), mental health (MH), role limitations due to emotional problems (RE), energy/vitality (VT), and social functioning (SF). The RP and RE scales have been modified in the veterans version from yes/no responses to five point ordinal choices. Otherwise the scale is comparable to the Medical Outcomes SF-36 functional assessment scale.
Veterans Quality of Life Assessment Scale (SF-36v) change from week 0 | 18 months
  Standardized, patient-rated cross-sectional scale measuring subjective physical and emotional health across 8 domains: general health (GH), physical function (PF), role limitations due to physical health (RP), bodily pain (BP), mental health (MH), role limitations due to emotional problems (RE), energy/vitality (VT), and social functioning (SF). The RP and RE scales have been modified in the veterans version from yes/no responses to five point ordinal choices. Otherwise the scale is comparable to the Medical Outcomes SF-36 functional assessment scale.
Veterans Quality of Life Assessment Scale (SF-36v) change from week 0 | 21 months
  Standardized, patient-rated cross-sectional scale measuring subjective physical and emotional health across 8 domains: general health (GH), physical function (PF), role limitations due to physical health (RP), bodily pain (BP), mental health (MH), role limitations due to emotional problems (RE), energy/vitality (VT), and social functioning (SF). The RP and RE scales have been modified in the veterans version from yes/no responses to five point ordinal choices. Otherwise the scale is comparable to the Medical Outcomes SF-36 functional assessment scale.
Veterans Quality of Life Assessment Scale (SF-36v) change from week 0 | 24 months
  Standardized, patient-rated cross-sectional scale measuring subjective physical and emotional health across 8 domains: general health (GH), physical function (PF), role limitations due to physical health (RP), bodily pain (BP), mental health (MH), role limitations due to emotional problems (RE), energy/vitality (VT), and social functioning (SF). The RP and RE scales have been modified in the veterans version from yes/no responses to five point ordinal choices. Otherwise the scale is comparable to the Medical Outcomes SF-36 functional assessment scale.
Davidson Trauma Scale (DTS) change from week 0 | 3 months
  The DTS is a 17 item self rated scale with each item corresponding to the 17 DSM-IV-TR symptoms of PTSD. Those 17 items comprise 3 clusters: Intrusive, Avoidance/Numbing, and Hyperarousal. The severity and frequency of each symptom is rated along with the distress associated with those symptoms.
Davidson Trauma Scale (DTS) change from week 0 | 6 months
  The DTS is a 17 item self rated scale with each item corresponding to the 17 DSM-IV-TR symptoms of PTSD. Those 17 items comprise 3 clusters: Intrusive, Avoidance/Numbing, and Hyperarousal. The severity and frequency of each symptom is rated along with the distress associated with those symptoms.
Davidson Trauma Scale (DTS) change from week 0 | 9 months
  The DTS is a 17 item self rated scale with each item corresponding to the 17 DSM-IV-TR symptoms of PTSD. Those 17 items comprise 3 clusters: Intrusive, Avoidance/Numbing, and Hyperarousal. The severity and frequency of each symptom is rated along with the distress associated with those symptoms.
Davidson Trauma Scale (DTS) change from week 0 | 12 months
  The DTS is a 17 item self rated scale with each item corresponding to the 17 DSM-IV-TR symptoms of PTSD. Those 17 items comprise 3 clusters: Intrusive, Avoidance/Numbing, and Hyperarousal. The severity and frequency of each symptom is rated along with the distress associated with those symptoms.
Davidson Trauma Scale (DTS) change from week 0 | 15 months
  The DTS is a 17 item self rated scale with each item corresponding to the 17 DSM-IV-TR symptoms of PTSD. Those 17 items comprise 3 clusters: Intrusive, Avoidance/Numbing, and Hyperarousal. The severity and frequency of each symptom is rated along with the distress associated with those symptoms.
Davidson Trauma Scale (DTS) change from week 0 | 18 months
  The DTS is a 17 item self rated scale with each item corresponding to the 17 DSM-IV-TR symptoms of PTSD. Those 17 items comprise 3 clusters: Intrusive, Avoidance/Numbing, and Hyperarousal. The severity and frequency of each symptom is rated along with the distress associated with those symptoms.
Davidson Trauma Scale (DTS) change from week 0 | 21 months
  The DTS is a 17 item self rated scale with each item corresponding to the 17 DSM-IV-TR symptoms of PTSD. Those 17 items comprise 3 clusters: Intrusive, Avoidance/Numbing, and Hyperarousal. The severity and frequency of each symptom is rated along with the distress associated with those symptoms.
Davidson Trauma Scale (DTS) change from week 0 | 24 months
  The DTS is a 17 item self rated scale with each item corresponding to the 17 DSM-IV-TR symptoms of PTSD. Those 17 items comprise 3 clusters: Intrusive, Avoidance/Numbing, and Hyperarousal. The severity and frequency of each symptom is rated along with the distress associated with those symptoms.
Global Assessment of Functioning Scale (GAF) change from week 0 | 3 months
  Clinician-rated, overall assessment of functional capacity related to psychiatric diagnosis that forms Axis V of DSM-IV TR multiaxial diagnostic assessment. It is designed to rate overall psychological, social and occupational functioning, but does not include any physical or environmental impairments. The patient is rated at the end of a diagnostic interview on a single score scale of 1-100, with the scale being divided into ten ranges of functioning.
Global Assessment of Functioning Scale (GAF) change from week 0 | 6 months
  Clinician-rated, overall assessment of functional capacity related to psychiatric diagnosis that forms Axis V of DSM-IV TR multiaxial diagnostic assessment. It is designed to rate overall psychological, social and occupational functioning, but does not include any physical or environmental impairments. The patient is rated at the end of a diagnostic interview on a single score scale of 1-100, with the scale being divided into ten ranges of functioning.
Global Assessment of Functioning Scale (GAF) change from week 0 | 9 months
  Clinician-rated, overall assessment of functional capacity related to psychiatric diagnosis that forms Axis V of DSM-IV TR multiaxial diagnostic assessment. It is designed to rate overall psychological, social and occupational functioning, but does not include any physical or environmental impairments. The patient is rated at the end of a diagnostic interview on a single score scale of 1-100, with the scale being divided into ten ranges of functioning.
Global Assessment of Functioning Scale (GAF) change from week 0 | 12 months
  Clinician-rated, overall assessment of functional capacity related to psychiatric diagnosis that forms Axis V of DSM-IV TR multiaxial diagnostic assessment. It is designed to rate overall psychological, social and occupational functioning, but does not include any physical or environmental impairments. The patient is rated at the end of a diagnostic interview on a single score scale of 1-100, with the scale being divided into ten ranges of functioning.
Global Assessment of Functioning Scale (GAF) change from week 0 | 15 months
  Clinician-rated, overall assessment of functional capacity related to psychiatric diagnosis that forms Axis V of DSM-IV TR multiaxial diagnostic assessment. It is designed to rate overall psychological, social and occupational functioning, but does not include any physical or environmental impairments. The patient is rated at the end of a diagnostic interview on a single score scale of 1-100, with the scale being divided into ten ranges of functioning.
Global Assessment of Functioning Scale (GAF) change from week 0 | 18 months
  Clinician-rated, overall assessment of functional capacity related to psychiatric diagnosis that forms Axis V of DSM-IV TR multiaxial diagnostic assessment. It is designed to rate overall psychological, social and occupational functioning, but does not include any physical or environmental impairments. The patient is rated at the end of a diagnostic interview on a single score scale of 1-100, with the scale being divided into ten ranges of functioning.
Global Assessment of Functioning Scale (GAF) change from week 0 | 21 months
  Clinician-rated, overall assessment of functional capacity related to psychiatric diagnosis that forms Axis V of DSM-IV TR multiaxial diagnostic assessment. It is designed to rate overall psychological, social and occupational functioning, but does not include any physical or environmental impairments. The patient is rated at the end of a diagnostic interview on a single score scale of 1-100, with the scale being divided into ten ranges of functioning.
Global Assessment of Functioning Scale (GAF) change from week 0 | 24 months
  Clinician-rated, overall assessment of functional capacity related to psychiatric diagnosis that forms Axis V of DSM-IV TR multiaxial diagnostic assessment. It is designed to rate overall psychological, social and occupational functioning, but does not include any physical or environmental impairments. The patient is rated at the end of a diagnostic interview on a single score scale of 1-100, with the scale being divided into ten ranges of functioning.
Wechsler Adult Intelligence Scale III (WAIS-III)-Digit Span Subtest change from baseline | 6 months
  Standardized, two-part test of working memory consisting of digits forward, which measures subjects ability to repeat sequences of 3 to 9 digits; and digits backward in which subjects are asked to repeat two to eight numbers in reverse order.
Wechsler Adult Intelligence Scale III (WAIS-III)-Digit Span Subtest change from baseline | 24 months
  Standardized, two-part test of working memory consisting of digits forward, which measures subjects ability to repeat sequences of 3 to 9 digits; and digits backward in which subjects are asked to repeat two to eight numbers in reverse order.
Controlled Oral Word Association Test (COWAT) change from baseline | 6 months
  This test is a brief and sensitive measure of verbal association fluency and executive cognitive dysfunction. It measures the spontaneous production of words beginning with a given letter (phonetic association) or given class of words (semantic association) and the subjects are asked to produce as many words as possible within the time limits. F, A and S are the most commonly used letters and a common category is animals. Administration takes approximately 5-10 minutes.
Controlled Oral Word Association Test (COWAT) change from baseline | 24 months
  This test is a brief and sensitive measure of verbal association fluency and executive cognitive dysfunction. It measures the spontaneous production of words beginning with a given letter (phonetic association) or given class of words (semantic association) and the subjects are asked to produce as many words as possible within the time limits. F, A and S are the most commonly used letters and a common category is animals. Administration takes approximately 5-10 minutes.
The Clinician-Administered PTSD scale (CAPS) change from week 0 | 12 months
  This is a standardized structured, clinician administered interview that includes both questions confirming the diagnosis of PTSD (CAPSDx) as well as symptom severity over specified time periods (lifetime, past week or past month) based on the 17 symptoms of PTSD in DSM-III/II-R and IV across clusters of recurrence, avoidance/numbing and hyper-arousal symptoms (CAPS1-17 or CAPSSx).
Clinical Global Impression and Improvement Scales (CGI-S and CGI-I) change from week 0 | 10 months
  Standardized clinician-administered, cross-sectional assessment of global severity (CGI-S) of PTSD symptomatic status and improvement (CGI-I) from baseline on ordinal 7 point scale.
Ruff Figural Fluency Test (RFFT) change from baseline | 6 months
  This test measures the production of novel designs under time constraints and is intended to assess the capacity for fluid and divergent thinking, flexibility in shifting thinking, planning strategies and the ability to coordinate a process. Five dot stimuli are presented in 35 contiguous squares and subjects are asked to draw as many unique designs as possible by connecting the dots within each rectangle.
Ruff Figural Fluency Test (RFFT) change from baseline | 24 months
  This test measures the production of novel designs under time constraints and is intended to assess the capacity for fluid and divergent thinking, flexibility in shifting thinking, planning strategies and the ability to coordinate a process. Five dot stimuli are presented in 35 contiguous squares and subjects are asked to draw as many unique designs as possible by connecting the dots within each rectangle.
Hopkins Verbal Learning Test - Revised (HVLT-R) change from baseline | 6 months
  This test assesses immediate and delayed recall along with delayed recognition. The subject is provided 3 learning trials to remember an orally presented 12-word list (four nouns from each of 3 semantic categories). Following a 20-25 minute interval, delayed recall and yes/no recognition are assessed. The yes/no recognition is where subjects are also asked to identify the words from a word list (12 target words and 12 non-target words) that is presented verbally. The test takes about 15 minutes excluding the delay interval which is preferably filled with intervening visuospatial tasks. Administration time is approximately 5-10 minutes excluding the 25 minute delay.
Hopkins Verbal Learning Test - Revised (HVLT-R) change from baseline | 24 months
  This test assesses immediate and delayed recall along with delayed recognition. The subject is provided 3 learning trials to remember an orally presented 12-word list (four nouns from each of 3 semantic categories). Following a 20-25 minute interval, delayed recall and yes/no recognition are assessed. The yes/no recognition is where subjects are also asked to identify the words from a word list (12 target words and 12 non-target words) that is presented verbally. The test takes about 15 minutes excluding the delay interval which is preferably filled with intervening visuospatial tasks. Administration time is approximately 5-10 minutes excluding the 25 minute delay.
Brief Visual Memory Test - Revised (BVMT-R) change from baseline | 6 months
  This test is used to assess visual memory and consists of six alternate forms that give measures of recognition, rate of acquisition, immediate recall, and delayed recall. For 10 seconds, a subject is given a stimulus form consisting of six geometric figures in a 2 x 3 matrix. The tasks consist of immediately drawing as many of the figures as possible in their correct location and this task is repeated 25 minutes later. This is followed by a recognition trial in which the subject is asked to identify which six of the 12 presented figures were on the original form. About 15 minutes are required for the test, excluding the delay interval.
Brief Visual Memory Test - Revised (BVMT-R) change from baseline | 24 months
  This test is used to assess visual memory and consists of six alternate forms that give measures of recognition, rate of acquisition, immediate recall, and delayed recall. For 10 seconds, a subject is given a stimulus form consisting of six geometric figures in a 2 x 3 matrix. The tasks consist of immediately drawing as many of the figures as possible in their correct location and this task is repeated 25 minutes later. This is followed by a recognition trial in which the subject is asked to identify which six of the 12 presented figures were on the original form. About 15 minutes are required for the test, excluding the delay interval.
Boston Naming Test (BNT) change from baseline | 6 months
  The BNT assesses the ability to name pictured objects with 60 line drawings that are presented one at a time. Words range from common (tree) to low frequency/rare (abacus). Scores include number correct and the need for various types of cueing as two prompting cues are allowed (phonemic cue, stimulus cue). Scores can be compared with age-based norms. This test requires approximately 10-20 minutes.
Boston Naming Test (BNT) change from baseline | 24 months
  The BNT assesses the ability to name pictured objects with 60 line drawings that are presented one at a time. Words range from common (tree) to low frequency/rare (abacus). Scores include number correct and the need for various types of cueing as two prompting cues are allowed (phonemic cue, stimulus cue). Scores can be compared with age-based norms. This test requires approximately 10-20 minutes.
Hooper Visual Organization Test (VOT) change from baseline | 6 months
  This tests the ability of the subject to conceptually organize visual stimuli (pictures) that have been disarranged and allows the assessor to detect neurological impairment. The test consists of 30 line drawings of common objects that have been cut into pieces. These pieces are scattered and the task is to identify what the object would be if the pieces were put back correctly. Total test time is approximately 10-15 minutes.
Hooper Visual Organization Test (VOT) change from baseline | 24 months
  This tests the ability of the subject to conceptually organize visual stimuli (pictures) that have been disarranged and allows the assessor to detect neurological impairment. The test consists of 30 line drawings of common objects that have been cut into pieces. These pieces are scattered and the task is to identify what the object would be if the pieces were put back correctly. Total test time is approximately 10-15 minutes.
Rey-Osterrieth Complex Figure (CFT) change from baseline | 6 months
  The purpose of this test is to assess visuospatial perception, attention, planning, and visual and working memory, by the construction of a complex figure and then remembering it for later recall (3 minutes and a 30 minute delayed recall). Total test time is approximately 10-15 minutes, excluding the delay.
Rey-Osterrieth Complex Figure (CFT) change from baseline | 24 months
  The purpose of this test is to assess visuospatial perception, attention, planning, and visual and working memory, by the construction of a complex figure and then remembering it for later recall (3 minutes and a 30 minute delayed recall). Total test time is approximately 10-15 minutes, excluding the delay.
Clock Drawing Test change from baseline | 6 months
  This is a screening test for visuospatial and cognitive dysfunction. The subject is given an unlined sheet of paper and asked to construct a clock containing all the numbers and with the hands set to a specified time. Abnormal drawings can be a result of psychiatric conditions as well as other medical conditions. This test can be completed in about 5 minutes. Several standardized, quantitative scoring systems exist.
Clock Drawing Test change from baseline | 24 months
  This is a screening test for visuospatial and cognitive dysfunction. The subject is given an unlined sheet of paper and asked to construct a clock containing all the numbers and with the hands set to a specified time. Abnormal drawings can be a result of psychiatric conditions as well as other medical conditions. This test can be completed in about 5 minutes. Several standardized, quantitative scoring systems exist.
Wisconsin Card Sorting Test (WCST) change from baseline | 6 months
  This test measures the ability to form concepts, utilize feedback and "set-shift", which is the ability to display flexibility in the face of changing conditions. Four stimulus cards are placed in front of the subject who then is given two packs of response cards with 64 cards in each set. No instructions are given as to how to match the response cards to the stimulus - by color, design or quantity of symbols. Feedback is given each time a correct or incorrect selection is made. During the test the matching rules are altered and the subject must adjust by learning the new rules. The approximate time to complete this test is 15-30 minutes. Assesses dorsolateral prefrontal-subcortical circuit function
Wisconsin Card Sorting Test (WCST) change from baseline | 24 months
  This test measures the ability to form concepts, utilize feedback and "set-shift", which is the ability to display flexibility in the face of changing conditions. Four stimulus cards are placed in front of the subject who then is given two packs of response cards with 64 cards in each set. No instructions are given as to how to match the response cards to the stimulus - by color, design or quantity of symbols. Feedback is given each time a correct or incorrect selection is made. During the test the matching rules are altered and the subject must adjust by learning the new rules. The approximate time to complete this test is 15-30 minutes. Assesses dorsolateral prefrontal-subcortical circuit function
Stroop Color and Word Test (STROOP) change from baseline | 6 months
  This test is a measure of reaction time, selective attention, cognitive flexibility in terms of shifting perception to changing demands, and the ability to suppress a habitual response in favor of an unusual one. It is based upon the fact that we can read words faster than we can name colors. There are 3 parts to the test. In Part 1 (Color Reading), the subject has to read the word of the colors, (red, green, blue) which are printed either in black ink or in the color that corresponds to the printed word. In the Part 2 (Color Naming), the print color of the words does not correspond to the color name and the subject must name the printed word. In Part 3, the subject must name the color in which the color names are printed and disregard reading the word. An increased interference effect can occur in a variety of disorders which include mental disease. The entire test can be completed in about 5 minutes. Assesses dorsolateral prefrontal-subcortical circuit function
Stroop Color and Word Test (STROOP) change from baseline | 24 months
  This test is a measure of reaction time, selective attention, cognitive flexibility in terms of shifting perception to changing demands, and the ability to suppress a habitual response in favor of an unusual one. It is based upon the fact that we can read words faster than we can name colors. There are 3 parts to the test. In Part 1 (Color Reading), the subject has to read the word of the colors, (red, green, blue) which are printed either in black ink or in the color that corresponds to the printed word. In the Part 2 (Color Naming), the print color of the words does not correspond to the color name and the subject must name the printed word. In Part 3, the subject must name the color in which the color names are printed and disregard reading the word. An increased interference effect can occur in a variety of disorders which include mental disease. The entire test can be completed in about 5 minutes. Assesses dorsolateral prefrontal-subcortical circuit function
Iowa Gambling Task (IGT) change from baseline | 6 months
  This test simulates a real-life decision-making situation and assesses the subjects decision making under ambiguity as well as classifying the subjects decision-making behavior in terms of risk taking and risk aversion. Subjects are given 4 card decks with the goal of maximizing winnings. They are told that sometimes they will win and sometimes they will lose but they are not informed that 2 of the decks are "risky" because they are associated with large wins, but also large losses. It has been found that subjects with orbitofrontal cortex dysfunction continue to persevere with the risky decks.
Iowa Gambling Task (IGT) change from baseline | 24 months
  This test simulates a real-life decision-making situation and assesses the subjects decision making under ambiguity as well as classifying the subjects decision-making behavior in terms of risk taking and risk aversion. Subjects are given 4 card decks with the goal of maximizing winnings. They are told that sometimes they will win and sometimes they will lose but they are not informed that 2 of the decks are "risky" because they are associated with large wins, but also large losses. It has been found that subjects with orbitofrontal cortex dysfunction continue to persevere with the risky decks.
Mini Mental State Exam (MMSE) change from baseline | 6 months
  The purpose of this test is to provide a rapid "bedside" grade of severity of cognitive impairment. Over the course of approximately 10 minutes, it samples orientation, memory, concentration, language and visuospatial function via simple questions and problems. The maximum score is 30 and any score > 25 is considered to be normal functioning.
Mini Mental State Exam (MMSE) change from baseline | 24 months
  The purpose of this test is to provide a rapid "bedside" grade of severity of cognitive impairment. Over the course of approximately 10 minutes, it samples orientation, memory, concentration, language and visuospatial function via simple questions and problems. The maximum score is 30 and any score > 25 is considered to be normal functioning.
Change in PET CT 18-fluorodeoxyglucose metabolism from baseline | 15 months
  Pre-operatively, patients will undergo a provocative PET CT scan using fluorodeoxyglucose (FDG) assessing activity of the amygdalae, insulae and medial PFC regions. The provocation will consist of re-exposure of the patient to the initial trauma that caused PTSD using script-driven imagery as in prolonged exposure therapy. Baseline and 15 month scans will be compared both for resting and post-provocation metabolism. The hypothesis is that DBS reduces amygdala hyperactivity in PTSD patients. The PET CT scan data will be processed with a statistical parametric mapping method using SPM99 (Wellcome Department of Neurology, London, England). PET data in each voxel will be normalized and fitted in a linear statistical model. Hypotheses will be evaluated as contrasts where the linear compounds of the model parameters will be evaluated with t-tests transformed into a z-score. We will consider z>3.09 (P<0.001 one tail, uncorrected) as statistically significant.

OTHER OUTCOMES:
Life Function in PTSD Scale (LFIPS) change from week 0 | 1 month
  The LFIPS was developed specifically for this study as the current literature does not contain any standardized instruments that assess patient functioning from the perspective of a significant other. It consists of several operationalized measures in each of six domains: Family Life, Marriage, Leisure, Children, Social Interactions, and Work/Productivity. Each question is rated on a scale of 1-5 with 5=Excellent and 1=Terrible. Total scores range from 18-80 with a lower score indicative of poor life functioning.
Life Function in PTSD Scale (LFIPS) change from week 0 | 2 months
  The LFIPS was developed specifically for this study as the current literature does not contain any standardized instruments that assess patient functioning from the perspective of a significant other. It consists of several operationalized measures in each of six domains: Family Life, Marriage, Leisure, Children, Social Interactions, and Work/Productivity. Each question is rated on a scale of 1-5 with 5=Excellent and 1=Terrible. Total scores range from 18-80 with a lower score indicative of poor life functioning.
Life Function in PTSD Scale (LFIPS) change from week 0 | 3 months
  The LFIPS was developed specifically for this study as the current literature does not contain any standardized instruments that assess patient functioning from the perspective of a significant other. It consists of several operationalized measures in each of six domains: Family Life, Marriage, Leisure, Children, Social Interactions, and Work/Productivity. Each question is rated on a scale of 1-5 with 5=Excellent and 1=Terrible. Total scores range from 18-80 with a lower score indicative of poor life functioning.
Life Function in PTSD Scale (LFIPS) change from week 0 | 4 months
  The LFIPS was developed specifically for this study as the current literature does not contain any standardized instruments that assess patient functioning from the perspective of a significant other. It consists of several operationalized measures in each of six domains: Family Life, Marriage, Leisure, Children, Social Interactions, and Work/Productivity. Each question is rated on a scale of 1-5 with 5=Excellent and 1=Terrible. Total scores range from 18-80 with a lower score indicative of poor life functioning.
Life Function in PTSD Scale (LFIPS) change from week 0 | 5 months
  The LFIPS was developed specifically for this study as the current literature does not contain any standardized instruments that assess patient functioning from the perspective of a significant other. It consists of several operationalized measures in each of six domains: Family Life, Marriage, Leisure, Children, Social Interactions, and Work/Productivity. Each question is rated on a scale of 1-5 with 5=Excellent and 1=Terrible. Total scores range from 18-80 with a lower score indicative of poor life functioning.
Life Function in PTSD Scale (LFIPS) change from week 0 | 6 months
  The LFIPS was developed specifically for this study as the current literature does not contain any standardized instruments that assess patient functioning from the perspective of a significant other. It consists of several operationalized measures in each of six domains: Family Life, Marriage, Leisure, Children, Social Interactions, and Work/Productivity. Each question is rated on a scale of 1-5 with 5=Excellent and 1=Terrible. Total scores range from 18-80 with a lower score indicative of poor life functioning.
Life Function in PTSD Scale (LFIPS) change from week 0 | 7 months
  The LFIPS was developed specifically for this study as the current literature does not contain any standardized instruments that assess patient functioning from the perspective of a significant other. It consists of several operationalized measures in each of six domains: Family Life, Marriage, Leisure, Children, Social Interactions, and Work/Productivity. Each question is rated on a scale of 1-5 with 5=Excellent and 1=Terrible. Total scores range from 18-80 with a lower score indicative of poor life functioning.
Life Function in PTSD Scale (LFIPS) change from week 0 | 8 months
  The LFIPS was developed specifically for this study as the current literature does not contain any standardized instruments that assess patient functioning from the perspective of a significant other. It consists of several operationalized measures in each of six domains: Family Life, Marriage, Leisure, Children, Social Interactions, and Work/Productivity. Each question is rated on a scale of 1-5 with 5=Excellent and 1=Terrible. Total scores range from 18-80 with a lower score indicative of poor life functioning.
Life Function in PTSD Scale (LFIPS) change from week 0 | 9 months
  The LFIPS was developed specifically for this study as the current literature does not contain any standardized instruments that assess patient functioning from the perspective of a significant other. It consists of several operationalized measures in each of six domains: Family Life, Marriage, Leisure, Children, Social Interactions, and Work/Productivity. Each question is rated on a scale of 1-5 with 5=Excellent and 1=Terrible. Total scores range from 18-80 with a lower score indicative of poor life functioning.
Life Function in PTSD Scale (LFIPS) change from week 0 | 10 months
  The LFIPS was developed specifically for this study as the current literature does not contain any standardized instruments that assess patient functioning from the perspective of a significant other. It consists of several operationalized measures in each of six domains: Family Life, Marriage, Leisure, Children, Social Interactions, and Work/Productivity. Each question is rated on a scale of 1-5 with 5=Excellent and 1=Terrible. Total scores range from 18-80 with a lower score indicative of poor life functioning.
Life Function in PTSD Scale (LFIPS) change from week 0 | 11 months
  The LFIPS was developed specifically for this study as the current literature does not contain any standardized instruments that assess patient functioning from the perspective of a significant other. It consists of several operationalized measures in each of six domains: Family Life, Marriage, Leisure, Children, Social Interactions, and Work/Productivity. Each question is rated on a scale of 1-5 with 5=Excellent and 1=Terrible. Total scores range from 18-80 with a lower score indicative of poor life functioning.
Life Function in PTSD Scale (LFIPS) change from week 0 | 12 months
  The LFIPS was developed specifically for this study as the current literature does not contain any standardized instruments that assess patient functioning from the perspective of a significant other. It consists of several operationalized measures in each of six domains: Family Life, Marriage, Leisure, Children, Social Interactions, and Work/Productivity. Each question is rated on a scale of 1-5 with 5=Excellent and 1=Terrible. Total scores range from 18-80 with a lower score indicative of poor life functioning.
Life Function in PTSD Scale (LFIPS) change from week 0 | 13 months
  The LFIPS was developed specifically for this study as the current literature does not contain any standardized instruments that assess patient functioning from the perspective of a significant other. It consists of several operationalized measures in each of six domains: Family Life, Marriage, Leisure, Children, Social Interactions, and Work/Productivity. Each question is rated on a scale of 1-5 with 5=Excellent and 1=Terrible. Total scores range from 18-80 with a lower score indicative of poor life functioning.
Life Function in PTSD Scale (LFIPS) change from week 0 | 14 months
  The LFIPS was developed specifically for this study as the current literature does not contain any standardized instruments that assess patient functioning from the perspective of a significant other. It consists of several operationalized measures in each of six domains: Family Life, Marriage, Leisure, Children, Social Interactions, and Work/Productivity. Each question is rated on a scale of 1-5 with 5=Excellent and 1=Terrible. Total scores range from 18-80 with a lower score indicative of poor life functioning.
Life Function in PTSD Scale (LFIPS) change from week 0 | 15 months
  The LFIPS was developed specifically for this study as the current literature does not contain any standardized instruments that assess patient functioning from the perspective of a significant other. It consists of several operationalized measures in each of six domains: Family Life, Marriage, Leisure, Children, Social Interactions, and Work/Productivity. Each question is rated on a scale of 1-5 with 5=Excellent and 1=Terrible. Total scores range from 18-80 with a lower score indicative of poor life functioning.
Life Function in PTSD Scale (LFIPS) change from week 0 | 18 months
  The LFIPS was developed specifically for this study as the current literature does not contain any standardized instruments that assess patient functioning from the perspective of a significant other. It consists of several operationalized measures in each of six domains: Family Life, Marriage, Leisure, Children, Social Interactions, and Work/Productivity. Each question is rated on a scale of 1-5 with 5=Excellent and 1=Terrible. Total scores range from 18-80 with a lower score indicative of poor life functioning.
Life Function in PTSD Scale (LFIPS) change from week 0 | 21 months
  The LFIPS was developed specifically for this study as the current literature does not contain any standardized instruments that assess patient functioning from the perspective of a significant other. It consists of several operationalized measures in each of six domains: Family Life, Marriage, Leisure, Children, Social Interactions, and Work/Productivity. Each question is rated on a scale of 1-5 with 5=Excellent and 1=Terrible. Total scores range from 18-80 with a lower score indicative of poor life functioning.
Life Function in PTSD Scale (LFIPS) change from week 0 | 24 months
  The LFIPS was developed specifically for this study as the current literature does not contain any standardized instruments that assess patient functioning from the perspective of a significant other. It consists of several operationalized measures in each of six domains: Family Life, Marriage, Leisure, Children, Social Interactions, and Work/Productivity. Each question is rated on a scale of 1-5 with 5=Excellent and 1=Terrible. Total scores range from 18-80 with a lower score indicative of poor life functioning.
Amygdala DBS in posttraumatic stress disorder scale (ADIPS) change from baseline | Week 0
  This consists of 3 neuropsychological assessments and 1 symptom checklist. Standardized assessments are the Faux Pas test; International Affective Picture System from Center for the Study of Emotion and Attention (CSA) at National Institutes of Mental Health (NIMH); and the Facial Emotional Expression Recognition Test. The amygdala related behavioral changes checklist is a screening instrument developed for this study. It comprises 54 items divided into categories of personality, emotional, sensory, perceptual, behavioral and vegetative function. Each item is scored from -3 to +3 based on operationalized definitions of change from baseline. Total scores for each functional domain and the entire inventory may be calculated. It is designed to screen subjects for neuropsychiatric changes possibly associated with amygdala stimulation based on extensive review of clinical and research literature on the human amygdala.
Amygdala DBS in posttraumatic stress disorder scale (ADIPS) change from week 0 | 1 month
  This consists of 3 neuropsychological assessments and 1 symptom checklist. Standardized assessments are the Faux Pas test; International Affective Picture System from Center for the Study of Emotion and Attention (CSA) at National Institutes of Mental Health (NIMH); and the Facial Emotional Expression Recognition Test. The amygdala related behavioral changes checklist is a screening instrument developed for this study. It comprises 54 items divided into categories of personality, emotional, sensory, perceptual, behavioral and vegetative function. Each item is scored from -3 to +3 based on operationalized definitions of change from baseline. Total scores for each functional domain and the entire inventory may be calculated. It is designed to screen subjects for neuropsychiatric changes possibly associated with amygdala stimulation based on extensive review of clinical and research literature on the human amygdala.
Amygdala DBS in posttraumatic stress disorder scale (ADIPS) change from week 0 | 2 months
  This consists of 3 neuropsychological assessments and 1 symptom checklist. Standardized assessments are the Faux Pas test; International Affective Picture System from Center for the Study of Emotion and Attention (CSA) at National Institutes of Mental Health (NIMH); and the Facial Emotional Expression Recognition Test. The amygdala related behavioral changes checklist is a screening instrument developed for this study. It comprises 54 items divided into categories of personality, emotional, sensory, perceptual, behavioral and vegetative function. Each item is scored from -3 to +3 based on operationalized definitions of change from baseline. Total scores for each functional domain and the entire inventory may be calculated. It is designed to screen subjects for neuropsychiatric changes possibly associated with amygdala stimulation based on extensive review of clinical and research literature on the human amygdala.
Amygdala DBS in posttraumatic stress disorder scale (ADIPS) change from week 0 | 3 months
  This consists of 3 neuropsychological assessments and 1 symptom checklist. Standardized assessments are the Faux Pas test; International Affective Picture System from Center for the Study of Emotion and Attention (CSA) at National Institutes of Mental Health (NIMH); and the Facial Emotional Expression Recognition Test. The amygdala related behavioral changes checklist is a screening instrument developed for this study. It comprises 54 items divided into categories of personality, emotional, sensory, perceptual, behavioral and vegetative function. Each item is scored from -3 to +3 based on operationalized definitions of change from baseline. Total scores for each functional domain and the entire inventory may be calculated. It is designed to screen subjects for neuropsychiatric changes possibly associated with amygdala stimulation based on extensive review of clinical and research literature on the human amygdala.
Amygdala DBS in posttraumatic stress disorder scale (ADIPS) change from week 0 | 4 months
  This consists of 3 neuropsychological assessments and 1 symptom checklist. Standardized assessments are the Faux Pas test; International Affective Picture System from Center for the Study of Emotion and Attention (CSA) at National Institutes of Mental Health (NIMH); and the Facial Emotional Expression Recognition Test. The amygdala related behavioral changes checklist is a screening instrument developed for this study. It comprises 54 items divided into categories of personality, emotional, sensory, perceptual, behavioral and vegetative function. Each item is scored from -3 to +3 based on operationalized definitions of change from baseline. Total scores for each functional domain and the entire inventory may be calculated. It is designed to screen subjects for neuropsychiatric changes possibly associated with amygdala stimulation based on extensive review of clinical and research literature on the human amygdala.
Amygdala DBS in posttraumatic stress disorder scale (ADIPS) change from week 0 | 5 months
  This consists of 3 neuropsychological assessments and 1 symptom checklist. Standardized assessments are the Faux Pas test; International Affective Picture System from Center for the Study of Emotion and Attention (CSA) at National Institutes of Mental Health (NIMH); and the Facial Emotional Expression Recognition Test. The amygdala related behavioral changes checklist is a screening instrument developed for this study. It comprises 54 items divided into categories of personality, emotional, sensory, perceptual, behavioral and vegetative function. Each item is scored from -3 to +3 based on operationalized definitions of change from baseline. Total scores for each functional domain and the entire inventory may be calculated. It is designed to screen subjects for neuropsychiatric changes possibly associated with amygdala stimulation based on extensive review of clinical and research literature on the human amygdala.
Amygdala DBS in posttraumatic stress disorder scale (ADIPS) change from week 0 | 6 months
  This consists of 3 neuropsychological assessments and 1 symptom checklist. Standardized assessments are the Faux Pas test; International Affective Picture System from Center for the Study of Emotion and Attention (CSA) at National Institutes of Mental Health (NIMH); and the Facial Emotional Expression Recognition Test. The amygdala related behavioral changes checklist is a screening instrument developed for this study. It comprises 54 items divided into categories of personality, emotional, sensory, perceptual, behavioral and vegetative function. Each item is scored from -3 to +3 based on operationalized definitions of change from baseline. Total scores for each functional domain and the entire inventory may be calculated. It is designed to screen subjects for neuropsychiatric changes possibly associated with amygdala stimulation based on extensive review of clinical and research literature on the human amygdala.
Amygdala DBS in posttraumatic stress disorder scale (ADIPS) change from week 0 | 7 months
  This consists of 3 neuropsychological assessments and 1 symptom checklist. Standardized assessments are the Faux Pas test; International Affective Picture System from Center for the Study of Emotion and Attention (CSA) at National Institutes of Mental Health (NIMH); and the Facial Emotional Expression Recognition Test. The amygdala related behavioral changes checklist is a screening instrument developed for this study. It comprises 54 items divided into categories of personality, emotional, sensory, perceptual, behavioral and vegetative function. Each item is scored from -3 to +3 based on operationalized definitions of change from baseline. Total scores for each functional domain and the entire inventory may be calculated. It is designed to screen subjects for neuropsychiatric changes possibly associated with amygdala stimulation based on extensive review of clinical and research literature on the human amygdala.
Amygdala DBS in posttraumatic stress disorder scale (ADIPS) change from week 0 | 8 months
  This consists of 3 neuropsychological assessments and 1 symptom checklist. Standardized assessments are the Faux Pas test; International Affective Picture System from Center for the Study of Emotion and Attention (CSA) at National Institutes of Mental Health (NIMH); and the Facial Emotional Expression Recognition Test. The amygdala related behavioral changes checklist is a screening instrument developed for this study. It comprises 54 items divided into categories of personality, emotional, sensory, perceptual, behavioral and vegetative function. Each item is scored from -3 to +3 based on operationalized definitions of change from baseline. Total scores for each functional domain and the entire inventory may be calculated. It is designed to screen subjects for neuropsychiatric changes possibly associated with amygdala stimulation based on extensive review of clinical and research literature on the human amygdala.
Amygdala DBS in posttraumatic stress disorder scale (ADIPS) change from week 0 | 9 months
  This consists of 3 neuropsychological assessments and 1 symptom checklist. Standardized assessments are the Faux Pas test; International Affective Picture System from Center for the Study of Emotion and Attention (CSA) at National Institutes of Mental Health (NIMH); and the Facial Emotional Expression Recognition Test. The amygdala related behavioral changes checklist is a screening instrument developed for this study. It comprises 54 items divided into categories of personality, emotional, sensory, perceptual, behavioral and vegetative function. Each item is scored from -3 to +3 based on operationalized definitions of change from baseline. Total scores for each functional domain and the entire inventory may be calculated. It is designed to screen subjects for neuropsychiatric changes possibly associated with amygdala stimulation based on extensive review of clinical and research literature on the human amygdala.
Amygdala DBS in posttraumatic stress disorder scale (ADIPS) change from week 0 | 10 months
  This consists of 3 neuropsychological assessments and 1 symptom checklist. Standardized assessments are the Faux Pas test; International Affective Picture System from Center for the Study of Emotion and Attention (CSA) at National Institutes of Mental Health (NIMH); and the Facial Emotional Expression Recognition Test. The amygdala related behavioral changes checklist is a screening instrument developed for this study. It comprises 54 items divided into categories of personality, emotional, sensory, perceptual, behavioral and vegetative function. Each item is scored from -3 to +3 based on operationalized definitions of change from baseline. Total scores for each functional domain and the entire inventory may be calculated. It is designed to screen subjects for neuropsychiatric changes possibly associated with amygdala stimulation based on extensive review of clinical and research literature on the human amygdala.
Amygdala DBS in posttraumatic stress disorder scale (ADIPS) change from week 0 | 11 months
  This consists of 3 neuropsychological assessments and 1 symptom checklist. Standardized assessments are the Faux Pas test; International Affective Picture System from Center for the Study of Emotion and Attention (CSA) at National Institutes of Mental Health (NIMH); and the Facial Emotional Expression Recognition Test. The amygdala related behavioral changes checklist is a screening instrument developed for this study. It comprises 54 items divided into categories of personality, emotional, sensory, perceptual, behavioral and vegetative function. Each item is scored from -3 to +3 based on operationalized definitions of change from baseline. Total scores for each functional domain and the entire inventory may be calculated. It is designed to screen subjects for neuropsychiatric changes possibly associated with amygdala stimulation based on extensive review of clinical and research literature on the human amygdala.
Amygdala DBS in posttraumatic stress disorder scale (ADIPS) change from week 0 | 12 months
  This consists of 3 neuropsychological assessments and 1 symptom checklist. Standardized assessments are the Faux Pas test; International Affective Picture System from Center for the Study of Emotion and Attention (CSA) at National Institutes of Mental Health (NIMH); and the Facial Emotional Expression Recognition Test. The amygdala related behavioral changes checklist is a screening instrument developed for this study. It comprises 54 items divided into categories of personality, emotional, sensory, perceptual, behavioral and vegetative function. Each item is scored from -3 to +3 based on operationalized definitions of change from baseline. Total scores for each functional domain and the entire inventory may be calculated. It is designed to screen subjects for neuropsychiatric changes possibly associated with amygdala stimulation based on extensive review of clinical and research literature on the human amygdala.
Amygdala DBS in posttraumatic stress disorder scale (ADIPS) change from week 0 | 13 months
  This consists of 3 neuropsychological assessments and 1 symptom checklist. Standardized assessments are the Faux Pas test; International Affective Picture System from Center for the Study of Emotion and Attention (CSA) at National Institutes of Mental Health (NIMH); and the Facial Emotional Expression Recognition Test. The amygdala related behavioral changes checklist is a screening instrument developed for this study. It comprises 54 items divided into categories of personality, emotional, sensory, perceptual, behavioral and vegetative function. Each item is scored from -3 to +3 based on operationalized definitions of change from baseline. Total scores for each functional domain and the entire inventory may be calculated. It is designed to screen subjects for neuropsychiatric changes possibly associated with amygdala stimulation based on extensive review of clinical and research literature on the human amygdala.
Amygdala DBS in posttraumatic stress disorder scale (ADIPS) change from week 0 | 14 months
  This consists of 3 neuropsychological assessments and 1 symptom checklist. Standardized assessments are the Faux Pas test; International Affective Picture System from Center for the Study of Emotion and Attention (CSA) at National Institutes of Mental Health (NIMH); and the Facial Emotional Expression Recognition Test. The amygdala related behavioral changes checklist is a screening instrument developed for this study. It comprises 54 items divided into categories of personality, emotional, sensory, perceptual, behavioral and vegetative function. Each item is scored from -3 to +3 based on operationalized definitions of change from baseline. Total scores for each functional domain and the entire inventory may be calculated. It is designed to screen subjects for neuropsychiatric changes possibly associated with amygdala stimulation based on extensive review of clinical and research literature on the human amygdala.
Amygdala DBS in posttraumatic stress disorder scale (ADIPS) change from week 0 | 15 months
  This consists of 3 neuropsychological assessments and 1 symptom checklist. Standardized assessments are the Faux Pas test; International Affective Picture System from Center for the Study of Emotion and Attention (CSA) at National Institutes of Mental Health (NIMH); and the Facial Emotional Expression Recognition Test. The amygdala related behavioral changes checklist is a screening instrument developed for this study. It comprises 54 items divided into categories of personality, emotional, sensory, perceptual, behavioral and vegetative function. Each item is scored from -3 to +3 based on operationalized definitions of change from baseline. Total scores for each functional domain and the entire inventory may be calculated. It is designed to screen subjects for neuropsychiatric changes possibly associated with amygdala stimulation based on extensive review of clinical and research literature on the human amygdala.
Amygdala DBS in posttraumatic stress disorder scale (ADIPS) change from week 0 | 18 months
  This consists of 3 neuropsychological assessments and 1 symptom checklist. Standardized assessments are the Faux Pas test; International Affective Picture System from Center for the Study of Emotion and Attention (CSA) at National Institutes of Mental Health (NIMH); and the Facial Emotional Expression Recognition Test. The amygdala related behavioral changes checklist is a screening instrument developed for this study. It comprises 54 items divided into categories of personality, emotional, sensory, perceptual, behavioral and vegetative function. Each item is scored from -3 to +3 based on operationalized definitions of change from baseline. Total scores for each functional domain and the entire inventory may be calculated. It is designed to screen subjects for neuropsychiatric changes possibly associated with amygdala stimulation based on extensive review of clinical and research literature on the human amygdala.
Amygdala DBS in posttraumatic stress disorder scale (ADIPS) change from week 0 | 21 months
  This consists of 3 neuropsychological assessments and 1 symptom checklist. Standardized assessments are the Faux Pas test; International Affective Picture System from Center for the Study of Emotion and Attention (CSA) at National Institutes of Mental Health (NIMH); and the Facial Emotional Expression Recognition Test. The amygdala related behavioral changes checklist is a screening instrument developed for this study. It comprises 54 items divided into categories of personality, emotional, sensory, perceptual, behavioral and vegetative function. Each item is scored from -3 to +3 based on operationalized definitions of change from baseline. Total scores for each functional domain and the entire inventory may be calculated. It is designed to screen subjects for neuropsychiatric changes possibly associated with amygdala stimulation based on extensive review of clinical and research literature on the human amygdala.
Amygdala DBS in posttraumatic stress disorder scale (ADIPS) change from week 0 | 24 months
  This consists of 3 neuropsychological assessments and 1 symptom checklist. Standardized assessments are the Faux Pas test; International Affective Picture System from Center for the Study of Emotion and Attention (CSA) at National Institutes of Mental Health (NIMH); and the Facial Emotional Expression Recognition Test. The amygdala related behavioral changes checklist is a screening instrument developed for this study. It comprises 54 items divided into categories of personality, emotional, sensory, perceptual, behavioral and vegetative function. Each item is scored from -3 to +3 based on operationalized definitions of change from baseline. Total scores for each functional domain and the entire inventory may be calculated. It is designed to screen subjects for neuropsychiatric changes possibly associated with amygdala stimulation based on extensive review of clinical and research literature on the human amygdala.
Electroencephalographic (EEG) Telemetry Session | 3-4 weeks after surgery
  Before initiation of experimental stimulation, subjects will be admitted to the Neurology EEG Telemetry Unit to test stimulus parameters for 1) after-discharges placing patients at high risk of seizures; 2) changes in vital signs posing risk of adverse health outcomes; 3) Changes in cardiac rhythm on electrocardiogram (ECG); and 4) changes in behavior portending significant safety risk if they were to occur at home in an unsupervised setting. Initial stimulation will be at 2.5 V, 120 μs pulse width and 160 Hz frequency. Amplitude will then be increased progressively to a maximum of 7 V. Pulse width will then be increased to a maximum of 210 μs pulse width. Finally, frequency will then be increased to a maximum of 200 Hz. Side effects will be specifically noted throughout. If a serious side effect occurs, the last parameter changed will be kept at a maximum of 60 % of the threshold value during subsequent experimental stimulation, and other parameters will not be increased.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph J Koek, MD, Principal Investigator — VA Greater Los Angeles; Jean-Philippe Langevin, MD, Principal Investigator — Southern Arizona VA Healthcare System AND VA Greater Los Angeles
Locations (1):
- VA Greater Los Angeles Healthcare System, Los Angeles, California, United States

REFERENCES:
- [Background] Langevin JP. The amygdala as a target for behavior surgery. Surg Neurol Int. 2012;3(Suppl 1):S40-6. doi: 10.4103/2152-7806.91609. Epub 2012 Jan 14. PMID 22826810
- [Background] Langevin JP, De Salles AA, Kosoyan HP, Krahl SE. Deep brain stimulation of the amygdala alleviates post-traumatic stress disorder symptoms in a rat model. J Psychiatr Res. 2010 Dec;44(16):1241-5. doi: 10.1016/j.jpsychires.2010.04.022. Epub 2010 May 26. PMID 20537659